CLINICAL TRIAL: NCT00497510
Title: Feasibility Study of Short-Term Effects of Chiropractic Manipulation on Older Adults With Impaired Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-04052006
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Musculoskeletal Equilibrium
Keywords: Balance; Chiropractic; Older Adults
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Chiropractic manipulation

SUMMARY:
To study the effect of chiropractic care and a specific exercise program on balance in older adults.

DETAILED DESCRIPTION:
Fall prevention in older adults is a significant public health issue that all health care providers must address. At this time, chiropractors, the most commonly used complementary and alternative medicine (CAM) practitioners, have not been systematically involved in either interventions for or research related to fall prevention and risk factor reduction. However, it is possible that body-based CAM practitioners such as chiropractors might make important contributions to decreasing fall risk through affecting musculoskeletal function and managing chronic pain, factors which may affect balance, an important risk factor for falls.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or older
2. Able to stand steadily without assistance on one leg for no more than 5 seconds (determined by averaging the time for both legs)
3. Able to attend all scheduled sessions (by self-report.)

Exclusion Criteria:

1. Non-ambulatory (that is, wheelchair bound); this precludes required balance testing; however, potential patients requiring assistive devices such as canes and walkers are not excluded.
2. received chiropractic care, physical therapy or any other manual care procedure within the past three months (by self report)
3. began an exercise program targeting balance and/or lower body strength within past month (by self report)
4. contraindications to CMT or mild-exertion exercise, as determined by the clinician through physical exam and x-rays (if indicated). Contraindications included but are not limited to: unstable or severe medical condition; severe osteoporosis, fracture or other osseous abnormalities; "high cardiovascular risk", ie.e. persons with known cardiovascular, pulmonary or metabolic disease, or one or more major signs/symptoms suggestive of cardiovascular and pulmonary disease
5. absence of indications for CMT, as determined by the clinician through history, physical exam, orthopedic tests, and static and motion palpation. Indications for CMT include identification of decreased or increased joint mobility usually accompanied by tenderness and muscle tension and spasm.
6. unable to understand English or Spanish adequately to complete study forms and questionnaires, since for this study we do not have study personnel fluent in other languages.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Specific Aim 1: Recruitment Tracking | through July 2007
Completeness of calendar collection, comparisons of baseline characteristics and assessments, qualitative assessment of utility of surveillance procedures. | Through July 2007
Documentation of Clinic Personnel Skills | Through July 2007
Statistical Analysis | Through July 2007

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hawk, DC, PhD., Principal Investigator — Cleveland Chiropractic College
Locations (2):
- United States (2):
  - Cleveland Chiropractic College Health Center, Kansas City, Missouri
  - Cleveland Chiropractic College, Kansas City, Missouri